CLINICAL TRIAL: NCT04822662
Title: The Effectiveness of The Education Program Based on The Individual and Family Self Management Theory Given For Epilepsy Adolescents and Parents: Randomized Controlled Trial
Brief Title: The Individual and Family Self Management Theory Based Epilepsy Education Program's Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hilal Kurt, Lecturer, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayUh01
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Self Management; Epilepsy; Seizure; Quality of Life
Keywords: Epilepsy; Self-Management; Chronic Disease; Adolescent; Education
MeSH Terms: conditions — Epilepsy; Chronic Disease

STUDY DESIGN:
Intervention Model Description: In this study, stratified sampling was employed based on age and sex. Two strata, [12-14 age, girl] and [15-18 age, boy], were generated to ensure even distribution in terms of age and sex in each group. First, thirty-six adolescent were stratified into two groups (A and B), which were then stratified again into two: [12-14 age, girl] and [15-18 age, boy]. A scheme was developed to randomize the age and sex of [12-14, girl] and [15-18 age, boy] into two groups (A and B), resulting in the experimental and control groups stratified by the age and sex and blocked into paired-groups of (2:2/[12-14 age, girl]:[15-18 age, boy]). Permutation was also used to strike a balance between the strata. Block sets were generated for each combination of the prognostic factors (age and sex). The experimental and control groups were then randomized into the strata using a random numbers table.
Who Masked: Participant
Masking Description: Single Blinded (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Epilepsy education program (Experimental): The training prepared for epilepsy will be held in 3 main modules and 5 sessions with two weeks intervals. Each session will last 25 minutes. Trainings will be given to adolescents and their parents online.
  Interventions: Behavioral: Epilepsy Education Programme
- Control Group (No Intervention): The control group will receive standard epilepsy treatment without any training intervention. The group did not receive any other intervention.

INTERVENTIONS:
Behavioral: Epilepsy Education Programme — Firstly the Child Introduction Form and Parent Information Form were applied. Then the Child's Attitude Towards Self-Disease Scale, Seizure Self-Efficacy Scale for Children, Quality of Life Scale for Children were filled to children. Nurse-Parent Support Scale were applied to the parents in the Pretest and Post Test data.
  Arms: Experimental Group: Epilepsy education program

SUMMARY:
The aim of the study; to determine the effect of education program given to adolescents diagnosed with epilepsy and their parents based on Ryan and Sawin's individual and family self-management theory, on adolescents 'attitudes towards disease, self-efficacy, quality of life and parents' nurse-parent support levels.

DETAILED DESCRIPTION:
In addition to the expected effects of epilepsy on children, the course of the disease and the course of the child's life will change as the duration of life with the disease increases. In epilepsy, it is necessary to develop self-management behaviors in order to facilitate adaptation to the disease, to encourage seizure control and to increase the quality of life. Regular repetition of the trainings created within the framework of a certain plan to improve self-management behaviors is one of the recommended steps to strengthen the individual with chronic disease in the disease process. This randomized controlled study including aged 12-18 adolescents with a diagnosis of epilepsy, monotherapy, mental retardation without cerebral palsy, and no secondary disease and their parents. However, there isn't enough published research examining the effect of education program given to adolescents diagnosed with epilepsy and their parents based on Ryan and Sawin's individual and family self-management theory, on adolescents 'attitudes towards disease, self-efficacy, quality of life and parents' nurse-parent support levels.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of epilepsy for at least 6 months,
* Being in the age range of 12-18 years,
* Cerebral palsy, attention deficit, lack of mental retardation, except for a different physical or epilepsy,
* Receiving monotherapy treatment for epilepsy
* To be able to communicate in Turkish

Exclusion Criteria:

* Cerebral palsy, attention deficit, mental retardation other than epilepsy,
* Patients who are over the age of 18 or who switch to an adult care program,
* Not being open to communication and cooperation, not taking polytherapy
* Adolescents not continuing the monitoring phase or wanting to stop working at any stage,
* Prior history of seizures due to screen exposure

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Child Introduction Form | First measurement - Before education programme (1st week)
  The form consists of 15 questions that question the content dimension (risk factors specific to the disease, factors specific to the physical and social environment, individual and familial factors) and the process dimension concepts (disease-specific knowledge and beliefs, self-regulation, social facilitation).
Development of the Child Attitude Toward Illness Scale | First measurement - Before education programme (1st week)
  Child Attitude Toward Illness Scale was developed by Austin (1993) to measure the attitudes of children with chronic diseases towards their disease. The validity and reliability of the 13-item single-dimension scale was conducted by Ersun and Bolisik (2012) with children aged 9-17 years with epilepsy.
  The average score that can be obtained from the scale varies between 1 and 5. The average score of 1 and 2 indicates negative attitude, 3 indicates neutral attitude, 4 and 5 indicate positive attitude.
Seizure Self-Efficacy Scale for Children | First measurement - Before education programme (1st week)
  Seizure Self-efficacy Scale for Children was developed by Caplin et al. (2002) and adapted to Turkish by Tutar Güven and İşler Dalgıç (Tutar Güven and İsler 2015). It was conducted with children aged 9-18 years with epilepsy and the Cronbach's alpha value of the scale was 0.89. The scale consists of a single dimension with a 15-item five-point Likert structure and the scale items are scored between 1-5. indicates that it is.
The Children's Quality of Life Scale | First measurement - Before education programme (1st week)
  The Children's Quality of Life Scale was developed in 2001 by Varni et al. For adolescents aged 13-18. The internal consistency coefficient of the scale varies between 0.80-0.88. The Turkish validity and reliability study of the scale was conducted by Çakın Memik et al. In 2007 and the internal consistency coefficient was found to be 0.82. PedsQL, which is one of the general quality of life scales, is a quality of life scale suitable for use in both healthy and ill adolescents. It is a five-point Likert-type scale consisting of 23 items that determines the health-related quality of life of adolescents aged 13-18.
Parents Information Form | First measurement - Before education programme (1st week)
  This form was prepared by the researchers in line with the literature. In the form, the individual and self management theory consists of 15 questions regarding the concepts of content and process dimension.
Nurse-Parent Support Scale | First measurement - Before education programme (1st week)
  The Nurse Parent Support Scale, developed by Miles et al. (1999) and tested by Yigit et al in 2017, consists of 21 items in a five-point likert structure. There is no reverse item in the scale that measures perceived nurse support by parents. The scale consists of four sub-dimensions. The scale consists of four sub-dimensions. These; It consists of 21 items in total: "Information and Communication Support", "Emotional Support", "Respect Support", "Quality Care".

SECONDARY OUTCOMES:
Development of the Child Attitude Toward Illness Scale | Second measurement - After education programme (10th week)
  Development of the Child Attitude Toward Illness Scale was developed by Austin (1993) to measure the attitudes of children with chronic diseases towards their disease. The validity and reliability of the 13-item single-dimension scale was conducted by Ersun and Bolisik (2012) with children aged 9-17 years with epilepsy.
  The average score that can be obtained from the scale varies between 1 and 5. The average score of 1 and 2 indicates negative attitude, 3 indicates neutral attitude, 4 and 5 indicate positive attitude.
Seizure Self-Efficacy Scale for Children | Second measurement - After education programme (10th week)
  Seizure Self-efficacy Scale for Children was developed by Caplin et al. (2002) and adapted to Turkish by Tutar Güven and İşler Dalgıç (Tutar Güven and İsler 2015). It was conducted with children aged 9-18 years with epilepsy and the Cronbach's alpha value of the scale was 0.89. The scale consists of a single dimension with a 15-item five-point Likert structure and the scale items are scored between 1-5. indicates that it is.
The Children's Quality of Life Scale | Second measurement - After education programme (10th week)
  The Children's Quality of Life Scale was developed in 2001 by Varni et al. For adolescents aged 13-18. The internal consistency coefficient of the scale varies between 0.80-0.88. The Turkish validity and reliability study of the scale was conducted by Çakın Memik et al. In 2007 and the internal consistency coefficient was found to be 0.82. PedsQL, which is one of the general quality of life scales, is a quality of life scale suitable for use in both healthy and ill adolescents. It is a five-point Likert-type scale consisting of 23 items that determines the health-related quality of life of adolescents aged 13-18.
Nurse-Parent Support Scale | Second measurement - After education programme (10th week)
  The Nurse Parent Support Scale, developed by Miles et al. (1999) and tested by Yigit et al in 2017, consists of 21 items in a five-point likert structure. There is no reverse item in the scale that measures perceived nurse support by parents. The scale consists of four sub-dimensions. The scale consists of four sub-dimensions. These; It consists of 21 items in total: "Information and Communication Support", "Emotional Support", "Respect Support", "Quality Care".

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Kurt Sezer, Master, Principal Investigator — KTO Karatay University; Sibel KUCUKOGLU, Assoch prof, Study Director — Selcuk University; Abdullah Canbal, Dr, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Result] Austin JK, Huberty TJ. Development of the Child Attitude Toward Illness Scale. J Pediatr Psychol. 1993 Aug;18(4):467-80. doi: 10.1093/jpepsy/18.4.467. PMID 8410570
- [Result] Tutar Guven S, Isler A. Validity and Reliability of the Seizure Self-Efficacy Scale for Children with Epilepsy. Noro Psikiyatr Ars. 2015 Mar;52(1):47-53. doi: 10.5152/npa.2015.7399. Epub 2015 Mar 1. PMID 28360675
- [Result] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Result] Miles MS, Carlson J, Brunssen S. The nurse parent support tool. J Pediatr Nurs. 1999 Feb;14(1):44-50. doi: 10.1016/S0882-5963(99)80059-1. PMID 10063248
- [Result] Caplin D, Austin JK, Dunn DW, Shen J, Perkins S. Development of a self-efficacy scale for children and adolescents with epilepsy. Children's Health Care. 2002; 31(4): 295-309.
- [Result] Ersun A, Bolışık B. VALIDITY AND RELIABILITY OF THE TURKISH ADAPTATION OF THE CHILD ATTITUDE TOWARD ILLNESS SCALE. EGEHFD. 2012; 28:37-45.
- [Derived] Sezer HK, Kucukoglu S, Canbal A. The effectiveness of an individual and family self-management theory-based education program given for adolescents with epilepsy and parents: Randomized controlled trial. J Pediatr Nurs. 2024 Nov-Dec;79:171-180. doi: 10.1016/j.pedn.2024.08.026. Epub 2024 Sep 13. PMID 39276443